CLINICAL TRIAL: NCT01388244
Title: Risk-stratified Osteoporosis Strategy Evaluation Study (ROSE)
Acronym: ROSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: University of Southern Denmark (Other); University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Katrine Rubin, Professor, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: ROSE; S-20090127 (Other: The Ethics Comittee of the Region of Southern Denmark)
Record Dates: First submitted 2011-06-29; First posted 2011-07-06 (Estimated); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Osteoporosis
Keywords: Screening; Risk Assessment; Fractures; Absorptiometry, Photon; Fracture prevention; Women; Patient prespective
MeSH Terms: conditions — Osteoporosis; Fractures, Bone | interventions — Mass Screening; Absorptiometry, Photon

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Screening (Active Comparator): Two-step screening process using FRAX risk score assessment followed by DXA scanning for high risk participants.
  Interventions: Other: Screening
- Control (Other): Control arm - Fracture risk assessment by FRAX without any intervention
  Interventions: Other: Control

INTERVENTIONS:
Other: Screening — Screening by risk factor assessment (FRAX) followed by DXA
  Other Names: DXA scan
  Arms: Screening
Other: Control — Observation by use of register data
  Arms: Control

SUMMARY:
The Risk-stratified Osteoporosis Strategy Evaluation Study (ROSE) is a randomised population-based study, including 20,904 Danish women aged 65-80 years, investigating the effectiveness of a two-step screening programme for osteoporosis, using a questionnaire based on FRAX® followed by DXA-scan of those at highest risk. Further, the study is expected to provide knowledge about cost-effectiveness, patient preferences and acceptance of screening programme to prevent fractures

DETAILED DESCRIPTION:
Osteoporosis is highly prevalent especially in postmenopausal women. Approximately 46 % of all women will suffer at least one osteoporotic fracture after the age of 50. The US Preventive Services Task Force (USPSTF) and National Osteoporosis Foundation (NOF) recommend screening with dual-energy x-ray absorptiometry (DXA) in all women aged 65 years and above regardless of risk factors. Nevertheless, the use of clinical risk factors has been shown to enhance the risk-gradient and accuracy of fracture risk prediction. The FRAX risk assessment score was derived from large population-based cohorts and validated in separate validation cohorts. Its use as a risk assessment tool is endorsed by WHO, but no prospective studies examining the effect of a screening programme using a combination of FRAX and DXA in a two-step manner have been performed previously.

35,000 women aged 65-80 years were selected at random from the population in the Region of Southern Denmark and -before inclusion-randomised to either a screening group or a control group. As first step, a self- administered questionnaire regarding risk factors for osteoporosis based on FRAX® was issued to both groups. As second step, subjects in the screening group with a 10-year probability of major osteoporotic fractures ≥15 % were offered a DXA scan. Patients diagnosed with osteoporosis from the DXA scan were advised to see their GP and discuss pharmaceutical treatment according to Danish National guidelines.

The primary outcome is incident clinical fractures as evaluated through annual follow-up using the Danish National Patient Registry. The secondary outcomes are cost-effectiveness, participation rate and patient preferences. The aim of the ROSE study is to investigate the effectiveness of a two-step population based osteoporosis screening programme using FRAX® based on self-administered questionnaire to select women for DXA followed by the standard osteoporosis treatment according to national guidelines and delivered by GPs in the Region of Southern Denmark. Secondary aims are to clarify whether the screening programme is cost-effective and to assess the patients' preferences, experience and acceptance of the screening programme. Moreover, sub-studies allow assessment of the effectiveness of FRAX® alone or combined with individual clinical risk factors in the prediction of fractures and the impact of socioeconomic factors for participation and outcome.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Age 65-80 years
* Inhabitants of the Region of Southern Denmark

Exclusion Criteria:

* Self-reported use of antiosteoporotic treatment and a diagnose of osteoporosis
* Unability to give informed consent

Ages: 65 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 35000 (Actual)
Dates: Start 2010-02 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
The effect of screening for osteoporosis with a two-step programme involving FRAX risk score followed by DXA for the prevention of hip fracture and other osteoporosis-related fracture events | Three years follow-up on average
  Comparison of register data concerning hospitalizations for primarily hip fracture between the intervention and control group as a whole. Power calculations suggest three years of followup on average, but this time frame could be increased if participation falls short.

SECONDARY OUTCOMES:
Cost-effectiveness / cost-utility of a two-step screening programme. | Three years follow-up on average
  Comparison of register-based health related costs due to antiosteoporotic medications combined with generated costs due to hospitalizations for osteoporosis-related fractures. Follow-up time is defined by the primary outcome measure

CONTACTS AND LOCATIONS:
Overall Officials: Kim Brixen, Professor, Study Director — University og Southern Denmark, Odense University Hospital, Denmark
Locations (1):
- Dept. of Endocrinology, Odense University Hospital, Odense, Denmark

REFERENCES:
- [Result] Rubin KH, Holmberg T, Rothmann MJ, Hoiberg M, Barkmann R, Gram J, Hermann AP, Bech M, Rasmussen O, Gluer CC, Brixen K. The risk-stratified osteoporosis strategy evaluation study (ROSE): a randomized prospective population-based study. Design and baseline characteristics. Calcif Tissue Int. 2015 Feb;96(2):167-79. doi: 10.1007/s00223-014-9950-8. Epub 2015 Jan 13. PMID 25578146
- [Result] Rubin KH, Rothmann MJ, Holmberg T, Hoiberg M, Moller S, Barkmann R, Gluer CC, Hermann AP, Bech M, Gram J, Brixen K. Effectiveness of a two-step population-based osteoporosis screening program using FRAX: the randomized Risk-stratified Osteoporosis Strategy Evaluation (ROSE) study. Osteoporos Int. 2018 Mar;29(3):567-578. doi: 10.1007/s00198-017-4326-3. Epub 2017 Dec 7. PMID 29218381
- [Result] Holmberg T, Moller S, Rothmann MJ, Gram J, Herman AP, Brixen K, Tolstrup JS, Hoiberg M, Bech M, Rubin KH. Socioeconomic status and risk of osteoporotic fractures and the use of DXA scans: data from the Danish population-based ROSE study. Osteoporos Int. 2019 Feb;30(2):343-353. doi: 10.1007/s00198-018-4768-2. Epub 2018 Nov 21. PMID 30465216
- [Result] Hoiberg MP, Rubin KH, Holmberg T, Rothmann MJ, Moller S, Gram J, Bech M, Brixen K, Hermann AP. Use of antiosteoporotic medication in the Danish ROSE population-based screening study. Osteoporos Int. 2019 Jun;30(6):1223-1233. doi: 10.1007/s00198-019-04934-7. Epub 2019 Mar 26. PMID 30911782
- [Result] Rothmann MJ, Moller S, Holmberg T, Hojberg M, Gram J, Bech M, Brixen K, Hermann AP, Gluer CC, Barkmann R, Rubin KH. Non-participation in systematic screening for osteoporosis-the ROSE trial. Osteoporos Int. 2017 Dec;28(12):3389-3399. doi: 10.1007/s00198-017-4205-y. Epub 2017 Sep 5. PMID 28875257
- [Result] Rothmann MJ, Huniche L, Ammentorp J, Barkmann R, Gluer CC, Hermann AP. Women's perspectives and experiences on screening for osteoporosis (Risk-stratified Osteoporosis Strategy Evaluation, ROSE). Arch Osteoporos. 2014;9:192. doi: 10.1007/s11657-014-0192-1. Epub 2014 Aug 19. PMID 25134980
- [Result] Rothmann MJ, Ammentorp J, Bech M, Gram J, Rasmussen OW, Barkmann R, Gluer CC, Hermann AP. Self-perceived facture risk: factors underlying women's perception of risk for osteoporotic fractures: the Risk-Stratified Osteoporosis Strategy Evaluation study (ROSE). Osteoporos Int. 2015 Feb;26(2):689-97. doi: 10.1007/s00198-014-2936-6. Epub 2014 Nov 1. PMID 25361616
- [Derived] Petersen TG, Rubin KH, Javaid MK, Hermann AP, Akesson KE, Abrahamsen B. Long-term adherence to anti-osteoporosis medication and determinants of adherence in the population-based screening trial ROSE. Osteoporos Int. 2025 Apr;36(4):695-706. doi: 10.1007/s00198-025-07436-x. Epub 2025 Feb 24. PMID 39992408
- [Derived] Petersen TG, Abrahamsen B, Hoiberg M, Rothmann MJ, Holmberg T, Gram J, Bech M, Akesson KE, Javaid MK, Hermann AP, Rubin KH. Ten-year follow-up of fracture risk in a systematic population-based screening program: the risk-stratified osteoporosis strategy evaluation (ROSE) randomised trial. EClinicalMedicine. 2024 Apr 11;71:102584. doi: 10.1016/j.eclinm.2024.102584. eCollection 2024 May. PMID 38638398
- [Derived] Holmberg T, Bech M, Gram J, Hermann AP, Rubin KH, Brixen K. Point-of-Care Phalangeal Bone Mineral Density Measurement Can Reduce the Need of Dual-Energy X-Ray Absorptiometry Scanning in Danish Women at Risk of Fracture. Calcif Tissue Int. 2016 Mar;98(3):244-52. doi: 10.1007/s00223-015-0084-4. Epub 2015 Nov 21. PMID 26590810